CLINICAL TRIAL: NCT00738985
Title: Efficacy of Ezetimibe/Simvastatin 10/20 mg and MK0524A (1-2 g/Day) in Patients With Mixed Hyperlipidemia and Two or More Risk Factors to Cardiovascular Disease.
Brief Title: Efficacy of Ezetimibe/Simvastatin 10/20 mg and MK0524A (1-2 g/Day) in Mixed Hyperlipidemia and Two or More Risk Factors
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: The study was cancelled due to budget limitations
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Carlos A Aguilar Salinas, Instituto Nacional de Ciencias Medicas y Nutricion
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008_019
Record Dates: First submitted 2008-08-19; First posted 2008-08-21 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Cardiovascular Diseases; Hyperlipidemia
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias | interventions — Ezetimibe; Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ezetimibe/simvastatin 10/20 mg + placebo (Placebo Comparator): The intervention consisted of an isocaloric diet, an exercise program (30 min/day of aerobic activity) and ezetimibe (+) simvastatin 10/20 mg + placebo for 12 weeks. Safety and efficacy parameters are measured at baseline and 12 weeks later
  Interventions: Drug: ezetimibe/simvastatin 10/20 mg + placebo
- ezetimibe/simvastatin 10/20 mg + MK0524A (Active Comparator): The intervention consisted of an isocaloric diet, an exercise program (30 min/day of aerobic activity) and ezetimibe/simvastatin 10/20 mg + MK0524A 1 gr for 6 weeks, if efficacy achieved will continue with ezetimibe (+) simvastatin 10/20 mg + MK0524A 1 gr + placebo; if not achieved, will receive ezetimibe (+) simvastatin 10/20 mg + MK0524A 2 gr for 6 weeks.
  Interventions: Drug: ezetimibe/simvastatin 10/20 mg + MK0524A

INTERVENTIONS:
Drug: ezetimibe/simvastatin 10/20 mg + placebo — Patients will receive placebo (sugar tablets) for up to 22 weeks.
  Other Names: No other drug is used per protocol in this study arm
  Arms: ezetimibe/simvastatin 10/20 mg + placebo
Drug: ezetimibe/simvastatin 10/20 mg + MK0524A — ezetimibe (+) simvastatin 10/20 mg for 18 weeks. Tablets
  Other Names: Vytorin; MK0653A
  Arms: ezetimibe/simvastatin 10/20 mg + MK0524A

SUMMARY:
To measure the percentage of patients who achieve all the treatment lipid goals being treated with ezetimibe/simvastatin 10/20 with or without MK0524A (1-2 g/day).

DETAILED DESCRIPTION:
Patients will receive placebo for 4 weeks, then Vytorin 10/20 mg for 6 weeks, if efficacy of treatment is achieved, they will continue with Vytorin 10/20 mg + placebo for 12 more weeks, if not achieved, will receive Vytorin 10/20 mg + MK0524A 1 gr for 6 weeks, if efficacy achieved will continue with Vytorin 10/20 mg + MK0524A 1 gr + placebo; if not achieved, will receive Vytorin 10/20 mg + MK0524A 2 gr for 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patient Without Ischemic Cardiovascular Disease Who During The Treatment With Statin Have LDL-C <130 Mg/Dl at Visit 1 Or Within The 6 Month Period Before Visit 1

Exclusion criteria:

* The use of any other lipid lowering agent
* Life expectancy lower than a year.
* Any condition that may interfere with the adherence to the study protocol

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-11; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Lipid parameters efficacy comparing ezetimibe/simvastatin alone vs. ezetimibe/simvastatin plus MK0524A (CORDAPTIVE) | 18 Week(s)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC